CLINICAL TRIAL: NCT04116190
Title: Feasibility of Multidisciplinary Telerehabilitation in Patients With Stroke - a Pilot Study
Brief Title: A Multidisciplinary Telerehabilitation for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vetrea Terveys Oy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Aimo2019
Record Dates: First submitted 2019-06-28; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Stroke Sequelae
Keywords: rehabilitation; stroke
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Consecutive sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (TR) (Experimental): Shortened inpatient rehabilitation mixed with home-based telerehabilitation.
  Interventions: Behavioral: Telerehabilitation
- Conventional rehabilitation (CR) (Experimental): Traditional inpatient rehabilitation
  Interventions: Behavioral: Conventional inpatient rehabilitation

INTERVENTIONS:
Behavioral: Telerehabilitation — Short inpatient multidisciplinary rehabilitation followed by home-based telerehabilitation and a short evaluation period at the end of it.
  Arms: Telerehabilitation (TR)
Behavioral: Conventional inpatient rehabilitation — Multidisciplinary inpatient rehabilitation, no adjustments due to the study.
  Arms: Conventional rehabilitation (CR)

SUMMARY:
Objective: Evaluate the feasibility of a multidisciplinary telerehabilitation for chronic stroke patients.

Design: Chronic stroke patients eligible for multidisciplinary rehabilitation funded by the Social Insurance Institution were enrolled between September 2017 and March 2018 in a consecutive basis to receive a mixed program of inpatient rehabilitation and telerehabilitation in their homes or a traditional inpatient rehabilitation only.

Intervention: A rehabilitation course with a 3-day inpatient stay followed by an 8-week telerehabilitation period completed by 2-day evaluation stay in a rehab center. The control group received conventional multidisciplinary rehabilitation for two weeks in an inpatient setting.

Outcome and measures: Change in the Finnish version of Functional Status Questionnaire (FSQFin), the World Health Organization Quality of Life - Short version (WHOQOL-Bref), the Barthel Index, the Beck Depression Inventory (BDI21), and the Goal Attainment Scale (GAS) and a patient satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (6 months or more) patient living in home
* eligible to receive rehabilitation funded by the Social Insurance Institution (meets the criteria of chronic disability and need for rehabilitation)
* for intervention group: capable to use a personal computer and telecommunication

Exclusion Criteria:

* no access or capability to use a personal computer
* significant problems in hearing, seeing or understanding information related to the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Finnish version of the Functional Status Questionnaire (FSQfin) | 8 weeks
  Functional Status Questionnaire for evaluating self-management in home. Includes three dimensions: self-care, mobility and domestic life. Scale range for each dimension is 0-100 and higher scores indicate better outcome.

SECONDARY OUTCOMES:
World Health Organization Quality of Life - short version (WHOQOL-Bref) | 8 weeks
  Quality of life assessment. Includes four dimensions: physical health, psychological health, social relationships and environment. Scale range for each dimension is 0-100 and higher scores indicate better outcome.
Beck Depression Inventory (BDI 21) | 8 weeks
  The Beck Depression Inventory for mood assessment. Scale range is 0-63 and higher scores indicate worse outcome.
Barthel Index | 8 weeks
  for assessing need for help in basic activities of daily living. Scale range is 0-100 and higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kauko Pitkanen, PhD, Study Director — VetreaNeuron
Locations (1):
- Vetrea, Kuopio, Northern Savonia, Finland